CLINICAL TRIAL: NCT02303691
Title: Neural Dimensions of Attention Bias Modification for Transdiagnostic Anxiety
Brief Title: Attention Bias Modification for Transdiagnostic Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Price, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5K23MH100259 (NIH)
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; Anxiety Disorders
Keywords: anxiety; attention bias modification; computer
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Completer analyses focused on prediction of active ABM outcomes using neural measures. Control arm used for effect size comparisons.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized Attention Bias Modification (Experimental)
  Interventions: Behavioral: Attention Bias Modification
- Computerized Neutral Training (Sham Comparator)
  Interventions: Behavioral: Neutral Training

INTERVENTIONS:
Behavioral: Attention Bias Modification — Excessive attention to threat is theorized to be a critical contributor to chronic anxiety symptoms and related negative health consequences. Attention Bias Modification, which directly targets this mechanism, is a highly cost-effective intervention with growing empirical support for its potential efficacy in clinically anxious populations.
  Arms: Computerized Attention Bias Modification
Behavioral: Neutral Training — A control version of computerized attention training.
  Arms: Computerized Neutral Training

SUMMARY:
This project seeks to identify neural mechanisms underlying the tendency for anxious individuals to pay more attention to threatening information than to other types of information. A computerized treatment designed to train individuals to reduce their attention towards threat will be tested, with a focus on understanding the aspects of brain function that predict response to the treatment. This work could ultimately lead to the ability to treat anxiety more effectively by directly targeting the aspects of brain function that are altered in a given patient.

ELIGIBILITY:
Inclusion Criteria:

* Participants will:

  1. be between the ages of 18 and 55 years,
  2. score >45 on the Spielberger State-Trait Anxiety Inventory-trait form.
  3. score >=75th percentile on the World Health Organization Disability Assessment Schedule 2.0

Exclusion Criteria:

1. Current medication or Cognitive-Behavioral Therapy for anxiety or depression;
2. Failure to meet standard Magnetic Resonance Imaging (MRI) inclusion criteria: those who have cardiac pacemakers, neural pacemakers, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants, Intrauterine Devices, metal braces, or other metal objects in their body, especially in the eye. If the subject has any metal or implants in the body they must be deemed safe by the MRI Research Center's safety screening procedure prior to enrollment. Dental fillings do not present a problem. Plastic or removable dental appliances do not require exclusion. Pregnancy, determined by pregnancy tests on females.
3. currently suicidal or at risk for harm to self or others,
4. visual disturbance (<20/40 as per the Snellen test, corrective lenses allowed)
5. <6th grade reading level as per the Wide Range Achievement Test
6. presence of bipolar, psychotic, autism spectrum, substance dependence, or primary depressive disorder
7. positive urine drug test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
CAPS--Hypervigilance item | 1 month

SECONDARY OUTCOMES:
Mood and Anxiety Symptoms Questionnaire | 1 month
Mini International Neuropsychiatric Interview (MINI) | 1 month
Attentional bias towards threat (Performance-based assessment of attentional bias towards threat based on reaction times and eye tracking) | immediate
  Performance-based assessment of attentional bias towards threat based on reaction times and eye tracking
Penn State Worry Questionnaire | 1 month
Liebowitz Social Anxiety Scale | 1 month
World Health Organization Disability Assessment Scale (WHODAS) | 1 month
Speilberger State-Trait Anxiety Inventory | 1 month
Beck Anxiety Inventory | 1 month

OTHER OUTCOMES:
Functional Magnetic Resonance Imaging | 1 month
  (collected post-treatment in subsample of active arm only)
Pupillometry | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Department of Psychiatry, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Price RB, Cummings L, Gilchrist D, Graur S, Banihashemi L, Kuo SS, Siegle GJ. Towards personalized, brain-based behavioral intervention for transdiagnostic anxiety: Transient neural responses to negative images predict outcomes following a targeted computer-based intervention. J Consult Clin Psychol. 2018 Dec;86(12):1031-1045. doi: 10.1037/ccp0000309. PMID 30507228
- [Derived] Price RB, Brown V, Siegle GJ. Computational Modeling Applied to the Dot-Probe Task Yields Improved Reliability and Mechanistic Insights. Biol Psychiatry. 2019 Apr 1;85(7):606-612. doi: 10.1016/j.biopsych.2018.09.022. Epub 2018 Oct 5. PMID 30449531